CLINICAL TRIAL: NCT07103954
Title: Comparative Effects of McKenzie Exercises vs. Mulligan Mobilization on Pain, Craniovertebral Angle, Functional Disability in Text Neck Syndrome
Brief Title: MCKENZIE EXERCISES VERSUS MULLIGAN MOBILIZATION IN TEXT NECK SYNDROME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sana Allah dita
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-05

CONDITIONS: Neck Pain; Text Neck Posture; Text Neck Syndrome
Keywords: MCKENZIE EXERCISES; MULLIGAN MOBILIZATION; TEXT NECK SYNDROME
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In this study, the outcome assessor will be blinded of treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McKenzie Exercise plus CPT (Experimental): In this group, McKenzie exercises with conventional physical therapy.
  Interventions: Other: McKenzie Exercises plus Conventional Physical Therapy
- Mulligan Exercise plus CPT (Active Comparator): In this group, Mulligan mobilization with conventional physical therapy. The
  Interventions: Other: Mulligan Mobilization with Conventional Physical Therapy

INTERVENTIONS:
Other: McKenzie Exercises plus Conventional Physical Therapy — First of all conventional physical therapy is applied. For this we will use transcutaneous electrical nerve stimulation (TENS) and hot pack, positioned over the neck region, for 15-20 minutes. This will help in improving blood flow and increasing muscle activation.
  For McKenzie exercises, the participant will be in a comfortable sitting posture with proper back support. He will be asked to perform the following exercises:
  1. Retraction in supine and sitting positions
  2. Retraction with patient and therapist overpressure
  3. Retraction with extension and rotation
  4. Rotation with patient and therapist overpressure
  5. Lateral flexion
  6. Lateral flexion with patient and therapist overpressure • All these exercises will be done with a hold of one or two seconds and the movement is then repeated for five to six times.
  Arms: McKenzie Exercise plus CPT
Other: Mulligan Mobilization with Conventional Physical Therapy — First of all conventional physical therapy is applied. For this we will use transcutaneous electrical nerve stimulation (TENS) and hot pack, positioned over the neck region, for 15-20 minutes. This will help in improving blood flow and increasing muscle activation.
  The Mulligan mobilization, the patient will be seated in a comfortable position on a chair and the therapist stood behind to perform the mulligan mobilization. A gliding force will be applied by the therapist on the patient's spinous process or on the facet joint of the superior vertebra of the target segment for treatment. This gliding force will be maintained by the therapist. Then the patient will move his head towards the painful side (flexion, extension, rotation, and lateral flexion), and more pressure will be applied by the patient at the end of active movement. The Mulligan mobilization will be repeated 10 times for 3 sets.
  Arms: Mulligan Exercise plus CPT

SUMMARY:
Neck pain is an important public health issue that affects the whole population. Consequently, there is a significant decrease in the quality of work and life and can have a negative socioeconomic impact on both individuals and society. For the treatment of pain in the spine and extremities, especially the neck, the McKenzie method of mechanical diagnosis and therapy (MMDT) is a popular choice. Mulligan mobilization approach was found to be beneficial for both pain and functioning in individuals with mechanical neck discomfort.

DETAILED DESCRIPTION:
Text Neck Syndrome, commonly referred to as turtle neck posture, is the fourth leading cause of disability globally. Different exercises and techniques have been implemented to manage it. Individually, there have been several studies conducted on McKenzie exercises and Mulligan mobilization. This study will provide valuable insights into the comparative effectiveness of McKenzie exercises and Mulligan mobilization for text neck syndrome. This study's findings will contribute to the development of evidence-based guidelines for managing TNS, enhancing clinical decision-making, and improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

Age 20 to 45 years

- Both genders will be included. A minimum of three hours must be spent using smartphones every day. More than one year of using any electronic gadgets. Craniovertebral Angle < 53

Exclusion Criteria:

* Any known illness that may cause pain in the upper limbs or neck.(e.g Rheumatoid arthritis) Any cervical spine injuries. Any neurological or cardiovascular issue (e.g epilepsy, hypertension) Pregnancy

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | The pain intensity will be measured using a visual analogue scale at baseline, and change in pain intensity will be measured at 2nd week and 4th week.
  The pain intensity will be measured using a visual analogue scale. The VAS is a self-reported scale that consists of anchor points for "no pain" and "worst possible pain" on a horizontal line (10 cm long). The patient is asked to mark at a single point along a 10-cm line that most accurately represent his level of pain. This line represents a continuum between the two ends of the scale, with "no pain" on the left end (0 cm) and "worst pain" on the right (10 cm).

SECONDARY OUTCOMES:
Functional disability | The functional disability will be measured at baseline, and change in function level will be measured at 2nd week and 4th week.
  It will be measured using the Neck Disability Index (NDI), which was the first instrument created to evaluate neck pain patients' self-rated disabilities. It consists of ten questions in the following domains: Pain Intensity, Personal Care, Lifting, Reading, Headaches, Concentration, Work, Driving, Sleeping, and Recreation. Each question contains six answer choices, scored from 0 (no disability) to 5 (complete disability). The scores for each section are then added. Scoring is reported on a 0-50 scale, 0 being the best possible score and 50 being the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Ashfaq Prof. Ahmad, PhD, Study Chair — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
In order to keep the privacy of participants and confidentiality.